CLINICAL TRIAL: NCT02871661
Title: Physical Therapy as Adjuvant Treatment of Vulvodynia: a Randomized Controled Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Marcela Grigol Bardin, Master in Obstetrics and Gynecology, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: State University of Campinas
Record Dates: First submitted 2016-07-19; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Vulvodynia
Keywords: vulvodynia; pelvic floor muscles; kinesiotherapy; electrical therapy; physical therapy; amitriptyline; female sexual dysfunction.
MeSH Terms: conditions — Vulvodynia | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amitriptyline (Active Comparator): This group will be treated with medication alone (amitriptyline hydrochloride, 25 mg) for chronic vulvar pain (vulvodynia).
  Interventions: Drug: Amitriptyline
- Amitriptyline plus kinesiotherapy (Active Comparator): This group will be treated with medication (amitriptyline hydrochloride, 25 mg) plus pelvic floor exercises such as Kegel contractions and stretching of pelvic floor muscles with patients own hands.
  Interventions: Drug: Amitriptyline; Other: Kinesiotherapy
- Amitriptyline plus IC (Quark) (Active Comparator): This group will be treated with medication (amitriptyline hydrochloride, 25 mg) plus electrical stimulation with Interferential Current (manufacturer: Quark Medical; Model: Dualpex 961 - program number 42): two electrodes put into the perineal surface area emitting interferential current, once a week for twenty minutes each, for eight weeks long.
  Interventions: Drug: Amitriptyline; Device: IC (Quark)

INTERVENTIONS:
Drug: Amitriptyline — Volunteers will take 25 milligrams of this medication every day from their enrollment until completing eight weeks long.
  Other Names: Amitriptyline hydrochloride
Other: Kinesiotherapy — Volunteers will be taught to contract their pelvic floor muscles right before stretching it, following a home protocol, every day for eight weeks long.
  Other Names: Kegel exercises plus muscle stretch
  Arms: Amitriptyline plus kinesiotherapy
Device: IC (Quark) — Volunteers will visit physical therapy clinic once a week to receive twenty minutes of electrical stimulation with Interferential Current (Duapex 961 of Quark Medical manufacturer) in their perineal area, for eight weeks long.
  Other Names: interferential current, Dualpex 961 - Quark
  Arms: Amitriptyline plus IC (Quark)

SUMMARY:
INTRODUCTION: Vulvodynia (chronic vulvar pain in the absence of clinical findings) has a negative impact over quality of life in women with this diagnose. The existing treatments, however, are manifold but insufficient. This study aims to verify the effectiveness of kinesiotherapy and electrotherapy as adjuvant methods in the treatment of vulvodynia. METHODS: A single-blind randomized controlled trial will examine 58 women, divided into three treatment arms: use of tricyclic antidepressant alone (hydrochloride Amitriptyline), amitriptyline hydrochloride associated with pelvic floor muscle exercises and amitriptyline hydrochloride associated with electrotherapy (interferential current). Exclusion criteria are: presence of infections or genital cancers, chronic degenerative diseases; younger than 18 years, neurological disease that jeopardizes the contraction of the muscles of the pelvic floor, taking antidepressant drugs that have interaction with amitriptyline hydrochloride and being pacemakers use. The parameters analyzed before and after treatment will be: muscle volume of the anus elevator and perfusion of the pudendal artery obtained with 3D ultrasound, subjective pain in vaginal intercourse (visual analog scale), monthly frequency of vaginal intercourse, pain referred within vulvar touch on physical examination (swab test from zero to 10) and female sexual function (Female Sexual Function questionnaire - FSFI). There will be a follow up of subjective pain in vaginal intercourse and monthly frequency of vaginal intercourse obtained by telephone contact with the voluntary on one, six and twelve months after the end of interventions. The data will be analyzed using Chi-square test of Pearson, Fisher exact and Mann-Whitney. The beginning and end of treatment will be compared using the Wilcoxon test (related samples) and McNemar (effect of the intervention), considering statistical significance level of 5%. The software used is the statistical analysis software (SAS) - Release 9.1, SAS Institute, Cary, North Carolina, USA, 2002-2003 and Statistical Package for the Social Sciences (SPSS) -Release 17.0.

DETAILED DESCRIPTION:
GOALS

1. General Check the effectiveness of physical therapy applied to the pelvic floor muscles used as an adjunct to standard treatment (amitriptyline hydrochloride) on the improvement of symptoms of vulvodynia.
2. Specific

Check and compare in women with vulvodynia before and after being randomly assigned to three treatment arms (drug only drug associated with therapeutic exercise or medication associated with electrotherapy with CI):

* Pain during intercourse and during the swab test obtained by Visual Analogue Scale (VAS);
* The scores obtained in the questionnaire Female Sexual Function Index (FSFI);
* The change in the volume of puborectal, pubococcygeus and iliococcygeal muscles accessed through Tridimensional Ultrasound (US3D);
* The variation of the perfusion of the pelvic floor muscles by pudendal artery obtained by 3D ultrasound;
* The effectiveness of therapeutic exercise in the improvement of vulvar pain to test swab and sexual intercourse by penetration in women diagnosed with vulvodynia;
* The effectiveness of electrical therapy with interferential current in the improvement of vulvar pain to test swab and sexual intercourse by penetration of women diagnosed with vulvodynia;
* Compare the effectiveness of electrical therapy and kinesiotherapy in the improvement of vulvar pain;
* Compare the effectiveness of physical therapy as an adjunct to standard against standard treatment alone.

SUBJECTS AND METHODS:

1. Study design:

   clinical trial randomized controlled single-blind. Designed according to the CONSORT standards, pending completion of the project after approval by Brazil Platform for final implementation, scheduled for July 2016.
2. Sample size:

   To calculate the sample size, we sought in literature studies addressing the main variables to be analyzed in this study (FSFI score after physical therapy intervention and medication versus medication, change in visual analog pain scale before and after the intervention).

   The study whose design and statistical analysis were closer than we propose in this project was used to calculate the sample, and its purpose was to compare in women with vulvodynia, the improvement in pain using the VAS pain and sexual function index using the FSFI after undergoing sessions of transcutaneous electrical stimulation (TENS) (65).

   Assuming type II alpha error probability equal to 0.05 and study of power equal to 80%, and considering the average VAS score of 8 (± 3.4) and 2.2 (± 6.1), the sample size calculation estimated using the Small software Stata 13.1 was n = 16 for each group, totaling n = 48. However, as a study with follow-up two months and assuming loss of follow-up of 20% of the total number of the sample, we assume a sampling size n = 58.
3. Variables and concepts:

3.1 Independent Variables Vulvodynia Characterized by present or absent, it is diagnosed by the presence of vulvar pain sexual penetration or touch gynecological self-reported, burning to light touch in the lobby (swab test [13]) and erythema. It can be classified as localized or generalized.

3.2 Dependent Variables Muscle thickness - Measure cross the levator ani muscle given in millimeters, obtained by 3D US in three situations: rest, maximum voluntary contraction and Valsalva; Perfusion pudendal artery - blood flow of the pudendal artery, given in millimeters per square centimeters (mm / cm2) obtained by 3D US.

Pain referred to the swab test - referred pain to perform the swab test, playing with a swab certain points of the vulvar vestibule, pointed using the visual analog scale (VAS) ranging from zero to 10, where ten is the highest grade concerning the higher pain threshold.

Pain said the vaginal penetration - mean referred pain during sexual intercourse with vaginal penetration, pointed using the visual analog scale (VAS) ranging from zero to 10, where ten is the maximum note to higher pain threshold.

FSFI - female sexual function index, as measured by the score obtained by the self-administered questionnaire FSFI (Female Sexual Function Index), which proposes to evaluate women's sexual response in the areas: desire, arousal, vaginal lubrication, orgasm, sexual satisfaction and pain. Assesses the relative strength of each field of female sexual response and transform subjective measures in objective, quantifiable and analyzable data. Applied in therapeutic exercise before and after the program applied to the pelvic floor.

3.3 Control variables BMI: body mass index, obtained by dividing weight in kilograms by height in meters squared. Categorized to assess the degree of obesity of an individual, it is considered underweight when BMI <20; ideal weight BMI = 20 to 25; overweight BMI = 26 to 30; moderate obesity BMI = 31 to 35; severe obesity BMI = 36 to 40; Morbid obesity BMI = 41 to 50; super obesity BMI> 50.

Gestation: number of times the respondent became pregnant, including abortions until the day of the interview (self reported); Delivery type: delivery route number taken by the respondent to the day of the interview, self reported, classified as: C-section; Forceps, vaginal; Frequency of sex: number of sexual contacts per month in the last six months (self reported); Number of sexual partners: number of partners in the last six months (self reported); Frequency of physical activity: number of times a week practicing physical activity on average in the last six months (self reported); Type of physical activity: type of physical activity carried out in the last six months (self reported) classified as: (I) strengthening (weight training, pilates class, functional training), (II) aerobic (walking, running, swimming, cycling, wrestling) and / or (III) stretching (stretching classes, yoga); (IV) sedentary.

Symptoms or pelvic floor dysfunction signs: self reported complaint by the patient in relation to the perineum such as dyspareunia, dysuria, redness, cracking, itching, vaginal flatus, urinary incontinence, fecal incontinence.

Treatment for vulvodynia used before kinesiotherapy: techniques and previously tested therapies to reduce the nuisance caused by vulvodynia.

Drug name, time and amount of drugs administered during the period of participation in the survey.

3.4 Descriptive Variables Age: elapsed time in years from the date of birth and date of the first interview, said the participant. Given in ordinal numbers; Education: number of years of study referred to by the subject. Given in ordinal numbers; Marital status: marital status of the subject at the time of the study. Categorized in (I) with a steady partner and (II) without a professional occupation; Skin color: skin color referred to by the subject. Categorized into (I) White and (II) not white; Smoking: current smoking habit, self reported by the interviewee, considering the options (I) yes or (II) not; Contraceptive methods that are used by women in order to prevent conception, informed by the participant, categorized into (I) male or female condom, (II) oral hormonal pill, (III) injectable hormonal contraceptive (IV) ligation of the fallopian tubes (V) or levonorgestrel copper intrauterine device (VI) rhythm, (VII) withdrawal, (VIII) and vasectomy (IX) other;

Subject Selection

Women who attend the outpatient genital infections and sexuality and are diagnosed with vulvodynia will be invited to participate in this study. Will also be distributed informative pamphlets on chronic vulvar pain and the methodology of this research in specialized clinics vulvodynia, vulvodynia groups on the Internet and clinics where researchers involved in this study attend. Women who agree to participate in the study aged over 18 years old will be interviewed in order to meet the criteria for inclusion in the study (Appendix I). The evaluation will be scheduled in the center of comprehensive care to women's health of Unicamp (CAISM) in physiotherapy clinic to perform the steps of the research participation.

The volunteers will be randomized through a computer program in www.randomizer.org obtained in three treatment arms: only amitriptyline, amitriptyline combined with kinesiotherapy applied to the pelvic floor and electrical therapy associated with the amitriptyline.

ELIGIBILITY:
Inclusion Criteria:

* Having had previous vaginal penetration
* Accept to perform kinesiotherapy sessions or electrical therapy once a week for two months
* Accept using medication (Amitriptyline hydrochloride) during the treatment period

Exclusion Criteria:

* Being pregnant
* Using drugs that negatively interfere with the hydrochloride Amtriptilina (ANNEX II)
* Having cognitive or literacy difficulties that prevent the understanding of self answered questionnaires such Female Sexual Function Index (FSFI).
* Refusing to sign the Informed Consent
* Neuromuscular disorders that interfere on the proper contraction of the pelvic floor muscles
* Having decompensated chronic degenerative diseases (tuberculosis, AIDS, hepatitis, diabetes, etc.)
* Using pacemaker or having cardiac arrhythmia
* Taking antidepressant monoamine oxidase inhibitor (MAOI) or Ayahuasca tea

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pain Scale Measurement | Eight weeks
  Effectiveness of the treatment for vulvodynia will be accessed through pain score scale from zero to ten, compared from day zero of treatment to day eight

SECONDARY OUTCOMES:
Female Sexual Index Function Improvement | Eight weeks
  Will be accessed through FSIF (Female Sexual Index Function questionnaire) score that goes from 2 to 36, compared from day zero of treatment to day eight, which indicates sexual disfunction pointed by scores below 26,55.
3D Ultrasound measurement of Pelvic Floor Muscle thickness and pudendal artery flow | Eight weeks
  A 3D Ultrassound will be used to access these outcomes and compare changes from day zero to day eight of treatment

OTHER OUTCOMES:
Interleukin 1-B Vaginal Inflammatory response | Eight weeks
  Vaginal fluid collected will be analysed in laboratory to access possible inflammatory response of vulva and vagina of women with vulvodynia obtained by comparing quantitatively interleukin 1-B presente before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paulo C Giraldo, MD, PhD, Study Director — University of Campinas, Brazil; Marcela G Bardin, PT, Master, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Unicamp, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goldstein AT, Pukall CF, Brown C, Bergeron S, Stein A, Kellogg-Spadt S. Vulvodynia: Assessment and Treatment. J Sex Med. 2016 Apr;13(4):572-90. doi: 10.1016/j.jsxm.2016.01.020. Epub 2016 Mar 25. PMID 27045258
- [Result] Reed BD, Caron AM, Gorenflo DW, Haefner HK. Treatment of vulvodynia with tricyclic antidepressants: efficacy and associated factors. J Low Genit Tract Dis. 2006 Oct;10(4):245-51. doi: 10.1097/01.lgt.0000225899.75207.0a. PMID 17012991
- [Result] Correa JB, Costa LO, Oliveira NT, Lima WP, Sluka KA, Liebano RE. Effects of the carrier frequency of interferential current on pain modulation and central hypersensitivity in people with chronic nonspecific low back pain: A randomized placebo-controlled trial. Eur J Pain. 2016 Nov;20(10):1653-1666. doi: 10.1002/ejp.889. Epub 2016 May 6. PMID 27150263
- [Result] Gentilcore-Saulnier E, McLean L, Goldfinger C, Pukall CF, Chamberlain S. Pelvic floor muscle assessment outcomes in women with and without provoked vestibulodynia and the impact of a physical therapy program. J Sex Med. 2010 Feb;7(2 Pt 2):1003-22. doi: 10.1111/j.1743-6109.2009.01642.x. Epub 2010 Jan 6. PMID 20059663
- [Result] Dionisi B, Anglana F, Inghirami P, Lippa P, Senatori R. [Use of transcutaneous electrical stimulation and biofeedback for the treatment of vulvodynia (vulvar vestibular syndrome): result of 3 years of experience]. Minerva Ginecol. 2008 Dec;60(6):485-91. Italian. PMID 18981976
- [Derived] Bardin MG, Giraldo PC, Fante JF, Carvalho de Araujo C, Cyr MP, Marques AA. Current Practices in Brazil on Diagnosis and Management of Women With Vulvodynia. J Low Genit Tract Dis. 2023 Apr 1;27(2):173-179. doi: 10.1097/LGT.0000000000000695. Epub 2023 Mar 3. PMID 36951987